CLINICAL TRIAL: NCT03443622
Title: Phase I Open-Label Dose-Escalating Study to Determine the Safety, Tolerability, Maximum Tolerated Dose, and Pharmacokinetics of SC-43 Oral Solution in Subjects With Refractory Solid Tumors
Brief Title: Phase I Study of SC-43 Oral Solution in Subjects With Refractory Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Another study has been started in other country.
Sponsor: SupremeCure Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SC-43-01
Record Dates: First submitted 2018-02-07; First posted 2018-02-23 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Refractory Solid Tumor
Keywords: SC-43; refractory solid tumor; Phase I

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- SC-43 100 mg/day (Experimental): SC-43 Oral Solution (100 mg/ml), 1 ml by mouth, q.d. for 28 days
  Interventions: Drug: SC-43 Oral Solution
- SC-43 200 mg/day (Experimental): SC-43 Oral Solution (100 mg/ml), 2 ml by mouth, q.d. for 28 days
  Interventions: Drug: SC-43 Oral Solution
- SC-43 400 mg/day (Experimental): SC-43 Oral Solution (100 mg/ml), 4 ml by mouth, q.d. for 28 days
  Interventions: Drug: SC-43 Oral Solution
- SC-43 600 mg/day (Experimental): SC-43 Oral Solution (100 mg/ml), 6 ml by mouth, q.d. for 28 days
  Interventions: Drug: SC-43 Oral Solution
- SC-43 900 mg/day (Experimental): SC-43 Oral Solution (100 mg/ml), 9 ml by mouth, q.d. for 28 days
  Interventions: Drug: SC-43 Oral Solution
- SC-43 1200 mg/day (Experimental): SC-43 Oral Solution (100 mg/ml), 12 ml by mouth, q.d. for 28 days
  Interventions: Drug: SC-43 Oral Solution

INTERVENTIONS:
Drug: SC-43 Oral Solution — SC-43 Oral Solution has drug substance of 1-[4-chloro-3(trifluoromethyl)phenyl-3-[3-(4-cyanophenoxy)] urea, or SC-43. SC-43 inhibits tumor growth through the activation of Src homology region 2 domain-containing phosphatase-1 (SHP-1) and the repression of p-STAT3 signalings. As a result of STAT3 inhibition by SC-43 treatment, decreased cell viability and enhanced apoptosis have been observed in cancer cells. The anti-tumor activity of SC-43 was also investigated in a variety of xenograft tumor models. Administration of SC-43 provides the tumor-bearing animals survival benefits, including the reduction of tumor volume and prolonged lifespan. SC-43 has been proposed to be evaluated as an anticancer therapeutic in in subjects with refractory solid tumors in the phase I trial.

SUMMARY:
This phase I study will be conducted in an open-label, conventional 3+3 dose escalation design manner (for the first 28 days of dosing) followed by an extension period for subjects responsive to the study drug to continue dosing up to 52 weeks. This study is intended to assess the safety and efficacy of the investigational product (IP), SC-43 Oral Solution, in subjects with refractory solid tumors. Subjects who have diseases progressing unresponsive to the previous treatments or who have no standard treatments for their current diseases will be enrolled in this study once the eligibility is confirmed.

During the first 28 days, the study will be done in the conventional 3+3 design to determine the maximum tolerated dose (MTD) of SC-43 Oral Solution. The dose will be increased in a step-wise fashion from the initial dose of 100 mg/day to the dose of 200, 400, 600, 900, and 1200 mg/day. The pharmacokinetics (PK) of SC-43 will also be measured in this period.

The dose of SC-43 Oral Solution will be escalated to the subsequent cohorts when there is no dose-limiting toxicity (DLT) in 3 subjects or only one DLT in 6 subjects of the previous cohort, and it is recommended by Data and Safety Monitoring Board (DSMB). The safety results will be reviewed by DSMB after the last subject in the each cohort has finished the Visit 6 (Day 29), and DSMB will determine if it is safe to proceed to the next dose cohort.

Subjects who have finished the 28-day dose escalation period and with complete response (CR), partial response (PR), or stable disease (SD) will be eligible to enter the extension period and continue SC-43 Oral Solution therapy up to 52 weeks or until occurrence of unacceptable toxicity, withdrawn consent, disease progression, not receiving medical benefit as considered by investigators, loss of follow-up, or death, whichever comes first. For ethical and safety concerns, the dosage used in this extension period can be adjusted and different from the original dosage assignment. The actual dose of SC-43 Oral Solution, which must be confirmed safe, administered during this extension period will be at the investigator's discretion.

DETAILED DESCRIPTION:
SC-43, has been shown to enhance the activity of Src homology region 2 domain-containing phosphatase-1 (SHP-1), leading suppression of STAT3 phosphorylation and tumor growth inhibition. SC-43 enhances SHP-1 activity by impairing the association between the N-SH2 domain and the PTP domain of SHP-1, triggering a conformational change of SHP-1 and relieving its autoinhibition. SC-43 treatment leads to cancer cell death in multiple cancer cell lines. SC-43 also exhibits anti-cancer activity in a variety of nonclinical xenograft tumor models.

ELIGIBILITY:
Inclusion Criteria:

1. Either gender, aged 20 to 75 years old (inclusive; the legal age of consent majority is 20 years old in Taiwan)
2. Life expectancy ≥ 12 weeks
3. With histologically or cytologically confirmed solid tumor(s) that is refractory to standard treatments, or for which a standard therapy is not available or is no longer effective
4. With at least one measurable target lesion as measured by MRI or CT according to Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 criteria
5. Subject who has received local therapies (such as surgery, radiation therapy, hepatic arterial embolization, or chemoembolization) is eligible. Local therapies must be completed at least 4 weeks prior to the baseline scan. However, the local therapy-treated tumor should be excluded for evaluation.
6. Eastern Cooperative Oncology Group (ECOG) performance status ≦2
7. If female subject or female spouse/partner of male subject is of childbearing potential, she/he must agree to use highly effective contraceptives from signing informed consent to 28 days after the last dose of study drug administration.

   At least two forms of birth control must be adopted and one of which must be a barrier method. Acceptable forms include:
   * Established use of oral, injected or implanted hormonal methods of contraception
   * Placement of an intrauterine device (IUD) or intrauterine system (IUS)
   * Barrier methods of contraception: condom, or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository
8. Dated and signed informed consent

Exclusion Criteria:

1. With primary central nervous system (CNS) malignancies or clinically active CNS metastases
2. The target solid tumor is lymphoma
3. Any of the following hematologic abnormalities:

   1. Hemoglobin < 8.0 g/dL
   2. Absolute neutrophil count (ANC) < 1,000/μL
   3. Platelets < 80,000 /μL
4. Any of the following serum chemistry abnormalities:

   1. Total bilirubin > 1.5 × ULN
   2. AST or ALT > 2.5 × ULN (> 5 × ULN in patients with HCC)
   3. γ-GT > 2.5 × ULN (> 5 × ULN in patients with HCC)
   4. ALP > 2.5 × ULN (> 5 × ULN in patients with HCC)
   5. Serum albumin < 2.5 g/dL
   6. Creatinine > 1.5 × ULN
   7. aPTT >1.5 × ULN
   8. INR >1.5 × ULN
   9. Any other ≥ Grade 3 (according to CTCAE v.5.0) laboratory abnormality at baseline (other than those listed above) Note: ULN = upper limit of normal; AST = aspartate transaminase; ALT = alanine transaminase; γ-GT = Gamma-glutamyl transferase; ALP = alkaline phosphatase; aPTT = activated partial thromboplastin time; INR = international normalized ratio of prothrombin time
5. History of organ or tissue transplantation
6. History of autoimmune disease
7. Active clinically serious infection
8. History of human immunodeficiency virus (HIV) infection
9. Significant cardiovascular disease, including:

   1. History of New York Heart Association (NYHA) class III or IV congestive heart failure
   2. Ongoing uncontrolled hypertension
   3. History of congenital long QT syndrome
   4. Ongoing prolonged corrected QT (QTc) interval defined as ≥ 450 msec
   5. History of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation)
10. With ascertained hypersensitivity to any ingredient of the investigational product or drugs with similar chemical structures, including sorafenib. If there is suspicion that the subject may have an allergy, the subject should be excluded.
11. Uncontrolled nausea or vomiting or any symptom that would prevent the ability to comply with daily oral SC-43 treatment
12. With significant gastrointestinal disorder(s) within 12 weeks prior to Screening that would, in the opinion of the investigator, prevent absorption of an orally available agent
13. Active bleeding during the last 4 weeks prior to Screening Visit
14. Requirement for ongoing immunosuppressive agents (including azathioprine, mycophenolate, cyclophosphamide, chlorambucil, methotrexate, cyclosporine), or systemic steroid with equivalent dosage higher than prednisolone 30 mg/day for more than 14 days
15. Received an investigational agent within 4 weeks prior to Screening
16. Had previous anti-cancer therapy (surgery, radiotherapy, chemotherapy, targeted therapy, immunotherapy, biology therapy, or hormonal therapy) within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to Screening Visit or has ongoing side effects (≥ Grade 2, according to CTCAE v.5.0) due to previously administered agents
17. Has undergone major surgery within 4 weeks before Screening Visit, or has elective or planned surgery to be conducted during the trial
18. Female with childbearing potential who has positive urine or serum pregnant test at Screening Visit or lactating
19. Is not considered to be suitable for this study, in the opinion of the investigator

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
maximum tolerated dose (MTD) | 28 days
  The highest dose level at which < 2 of 6 subjects experienced a dose limiting toxicity during the first 28 days of the treatment period.

SECONDARY OUTCOMES:
Objective response rate (ORR) according to RECIST criteria version 1.1 | 28 days
  Objective response rate (ORR) is defined as the proportion of subjects with complete response (CR) or partial response (PR) as best overall response evaluated according to RECIST criteria version 1.1 on MRI or CT results.
Disease control rate (DCR) according to RECIST criteria version 1.1 | 28 days
  Disease control rate (DCR) is defined as the proportion of subjects with complete response (CR), partial response (PR), or stable disease (SD) as best overall response evaluated according to RECIST criteria version 1.1 on MRI or CT results.
The maximum plasma concentration (Cmax) | 28 days
  PK blood samples will be collected at predefined time intervals, and the maximum plasma concentration will be determined.
Area under the plasma concentration versus time curve (AUC) | 28 days
  PK blood samples will be collected at predefined time intervals, and the AUC from time 0 to the last time point will be calculated.
Number of patients with treatment-related adverse events (AEs) based on NCI-CTCAE version 5.0 | 28 days
  An adverse event (AE) means any untoward medical occurrence in a subject or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. All AEs will be assessed for severity based on NCI-CTCAE version 5.0.